CLINICAL TRIAL: NCT05972434
Title: A Single-Center, Open-Label Safety-in-Use Clinical Trial to Assess the Topical Tolerability and Efficacy in Improving Hydration, Skin Barrier Function, and Skin Tone Uniformity of Two Facial Sunscreens (IPs) Under Controlled and Normal Conditions of Use on the Face by Adult Participants
Brief Title: A Study of Two Facial Sunscreens to Assess Its Effect in Improving Hydration, Skin Barrier Function, and Skin Tone Uniformity Under Controlled and Normal Conditions of Use on the Face by Adult Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CCSSKA005284; CCSSKA005284 (Other: Johnson & Johnson Consumer Inc. (J&JCI))
Record Dates: First submitted 2023-06-30; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Sunscreen A (Experimental): Eligible study participants will receive a standard liquid soap to be used on the face and forearms for 3 full days for an initial washout period in place of their usual soap. On their next visit to site an amount of IP will be topically applied to malar on one side of the participant's face by a qualified technician and other side of face will remain without product application (used for control). Six areas will also be marked on inner side of participant's forearms, approximately 5 centimeter (cm) from cubital region. These areas will be randomized, with 1 area for control (without product application) and other 5 areas for product application, being each of them for 02 IPs (Facial Sunscreen A and Face Sunscreen B) and 3 benchmarks. The products will be applied topically only once in marked areas. Next, participants will use Facial Sunscreen A in normal conditions at home for 28 +/- 2 days and then make the last study visit to complete the final analysis.
  Interventions: Other: Sunscreen A
- Group 2: Sunscreen B (Experimental): Eligible study participants will receive a standard liquid soap to be used on the face for 3 full days for an initial washout period in place of their usual soap. On their next visit to the Site an amount of the IP will be topically applied to the malar on one side of the participants' face by a qualified technician and the other side of the face will remain without product application (used for control). On their next visit to the Site an amount of the IP will be topically applied to the malar on one side of the participants' face by a qualified technician and the other side of the face will remain without product application (used for control). From Visit 2 to visit 4 participants will use the IP (Face Sunscreen B) at home until 56 +/-2 days of use.
  Interventions: Other: Sunscreen B

INTERVENTIONS:
Other: Sunscreen A — Participants will apply sunscreen A topically.
  Arms: Group 1: Sunscreen A
Other: Sunscreen B — Participants will apply sunscreen B topically.
  Arms: Group 2: Sunscreen B

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of 02 facial sunscreens (investigational products [IPs]) under controlled and normal conditions of use on the face for 28 and 56 days, respectively. This study will consist of 2 groups a) Group 1: will assess the safety and efficacy of a facial sunscreen in improving skin hydration and barrier function, through 12h of single application on the face in comparison with the control area (other side of face) and on the forearm, comparing 02 IPs versus control area (no product application) and 03 benchmarks; and through use of the IP under normal conditions for 28 +/- 2 days on the face, with assessments by instrumental measurements of corneometry, transepidermal water loss, image capture (Colorface) and assessments of the efficacy perceived by the participant; b) Group 2: will evaluate the safety and efficacy of a facial sunscreen in improving skin hydration and barrier function, through 12h of single application on the face; and through use of IP under normal conditions for 28 +/- 2 days on the face, with assessments by instrumental measurements of corneometry, transepidermal water loss, imaging (Colorface) and assessments of the efficacy perceived by the participant; in addition to evaluating the improvement in uniformity of facial skin tone through the use of IP under normal conditions for 56 +/- 2 days, with assessments by image analysis (Colorface), dermatological clinical analyses (radiance and homogeneity of skin tone),assessments of perceived efficacy, and emotional testimony by the participant.

ELIGIBILITY:
Inclusion Criteria:

* Participants of any ethnicity according to IBGE criteria
* Generally in good health based on medical history reported by the participant
* Able to read, write, speak, and understand Portuguese
* Capacity to consent to participation in the study
* Fitzpatrick Skin Type I to IV
* Intact skin in the test region
* Specific for Group 1: Participants with dry skin on the forearms (Corneometer score of maximum 40 arbitrary units (a.u.) at initial measurement before application of the products
* Participants with a maximum facial corneometry value of 60 a.u. at the initial measurement before the application of the products
* Participants presenting recent and repetitive complaints of discomfort caused by dry skin on the face, such as: pining, itching, irritation, et cetra
* Specific for Group 2: Participants who present lack of homogeneity in the tone of the facial skin due to hyperchromia caused by sun spots, solar lentigo, post-inflammatory hyperpigmentation, ephelid and mild melasma (proven by Dermatologist)
* Specific for Group 2: Participants who present lack of radiance in the skin (proven by Dermatologist)
* Individual who has signed the informed consent document (ICD) and image disclosure consent term (IDCT)
* Concordance to adhere to the procedures and requirements of the study and to attend the Site on the day(s) and time(s) determined for the evaluations
* For male participants: agree to shave 24 hours before visit 1, 2 and 3

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skin care products including sunscreen
* Presents with a skin condition that may confound the study results (specifically psoriasis, eczema, active atopic dermatitis, active skin cancer)
* Presents with primary/secondary lesions on test sites (example. scars, ulcers, vesicles, tattoos)
* Report having Type 1 or Type 2 diabetes or taking insulin or another anti-diabetic medication: presents immunological insufficiency; Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including; Immunosuppressive or steroidal drugs within 60 days before Visit 1; Non-steroidal anti-inflammatory drugs within 5 days before Visit 1; Antihistamines within 14 days before Visit 1
* Participants who are currently using or have recently used any facial products containing active skin barrier replacement and intense moisturizing ingredients such as: urea, ceramides, hyaluronic acid, glycerin, butters and oils, within 2 months prior to the start of the study
* Participants who have used cosmetic products for facial and body moisturizing (on the forearms) within 07 days prior to the start of the study
* Specific for Group 2: Participants who are using or have recently used any facial products containing active ingredients against spots: alpha or beta hydroxy acids (including salicylic acid), polyhydroxy acids, topical products containing retinol or retinol derivatives, hydroquinones, arbutin, niacinamide, N-acetylglucosamine, Thiamidol, kojic acid, azelaic acid, licorice extract, whitening peptides, vitamin C, or any other product capable of interfering with the uniformity of skin tone/spots, within 2 months prior to the start of the study
* Participants who have undergone invasive cosmetic or dermatological treatment in the test areas within 2 months prior to the start of the study or during the study
* Participants who are using any medication to treat diseases of the face or body
* Other diseases or medications that may directly interfere with the study or endanger the health of the research participant
* Is self-reported to be pregnant or planning to become pregnant during the study
* Has a history of or a concurrent health/other condition/situation which, in the opinion of the Study Physician, may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study
* Is simultaneously participating in any other study
* Is an employee/contractor or immediate family member of the principal investigator (PI), Study Site, or Sponsor
* Presents excessive hair in the evaluation regions that may interfere with the instrumental measurements. In the case of men, they will be instructed to shave 24 hours before the visit

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-06-23 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Groups 1 and 2: Skin Hydration as Assessed Through Instrumental Corneometry Measurements During 12 Hours of Visit 2 | 0 hour, 2 hours, 4 hours, 6 hours, 8 hours and 12 hours (Visit 2)
  Instrumental corneometry will be used to assess improvement in skin hydration during 12 hours of single application on one side of the face (hemi-face), in comparison with the control area (other side of face, without product application). The investigational product (IP) will be applied only once on half face, on the malar region, by a trained technician. The treated area and the control area will be tested in triplicate at each experimental time (T0h, T2h, T4h, T6h, T8h and T12h), with the corneometer instrument.
Groups 1 and 2: Skin Hydration as Assessed Through Instrumental Skin Corneometry Measurements at Day 28 +/- 2 | Up to Day 28 +/- 2
  Instrumental corneometry measurements will be used to assess improvement in skin hydration at Day 28 +/- 2 of application on the face (normal conditions of use). The IP will be applied on the entire face throughout the 28 days period. There should not be any type of product applied to the evaluation area at the time of the measurements.
Groups 1 and 2: Skin Barrier Integrity as Assessed Through Tewameter Measurements | Day 28 +/- 2
  Skin barrier measurements (an initial measurement at Visit 2 and a final measurement at Visit 3) will be performed with the Tewameter. A single transepidermal water loss (TEWL) measurement will be taken in the nasegenian region, on the face of the participants. There should not be any type of product applied to the evaluation area at the time of the measurements.
Groups 1 and 2: Participant's Self-perceived Efficacy Questionnaire to Assess Clinical Effectiveness | Day 28 +/- 2
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen will be reported. It is a 9-item questionnaire and each item is rated as totally disagree, disagree, neither agree nor disagree, agree and totally agree. Participants will additionally answer 1 question and rate it as liked very much, liked slightly, neither liked nor disliked, disliked slightly and disliked very much.
Group 1:Percentage of Participants with Adverse Events | Up to 28 +/- 2 days
  Percentage of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/ frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.
Group 2: Facial Skin Tone as Assessed Through Radiance/Brightness/Luminousness Scale | Up to Day 56 +/- 2
  To evaluate the parameters of radiance of the participant's skin tone, radiance/brightness/luminousness ordinal scale developed by the study site will be used. Radiance/Brightness/Luminousness scale is a 10-point system (0 to 9) that grades the intensity of these attributes, where 0 to 3: characteristic of "radiant, bright and luminous appearance" skin, 4 to 6: moderately radiant, and 7 to 9: characteristic of "dull/matte and/or pale" skin.
Group 2: Facial Skin Tone as Assessed Through Skin Tone Uniformity/Homogeneity Scale | Up to Day 56 +/- 2
  To evaluate the parameters of uniformity of the participant's skin tone, skin tone uniformity/homogeneity ordinal scale developed by the study site will be used. Skin tone uniformity/homogeneity ordinal scale is a 10-point system (0 to 9) that rates the intensity of these attributes, where 0 to 3 is characteristic of " even/healthy color" skin, 4 to 6 is moderately even, and 7 to 9 is characteristic of " irregular, discolored, spotted" skin.
Group 2: Facial Skin Tone as Assessed Through Image Analysis via Colorface | Day 56 +/- 2
  Image analysis via Colorface will be used to assess improvement in facial skin tone. The images of the participants faces will be captured with Colorface equipment (Newtone Technology) that will be operated by a trained technician.
Group 2: Testimonial Regarding the Experience with Sunscreen | Day 56
  A testimonial regarding the experience with sunscreen will be provided by the participants through an open question at the end of the study. The purpose is to know their opinion and experience using this product during the study.
Group 2:Percentage of Participants with Adverse Events | Up to 56 +/- 2 days
  Percentage of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/ frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.
Group 2: Participant's Self-perceived Efficacy Questionnaire to Assess Clinical Effectiveness | Day 56 +/-2
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 56 will be reported. Participants will answer 12 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree. Participants will additionally answer 2 questions and rate them as liked very much, liked slightly, neither liked nor disliked.

SECONDARY OUTCOMES:
Group 1 and 2: Skin Hydration as Assessed by Hydration Map | Up to Day 28+/- 2 days
  Facial images will be captured with ColorFace (Newtone Technology) equipment at the baseline and Day 28 to build a facial hydration map for the in-use study.
Group 1: Skin Hydration as Assessed Through Instrumental Forearms Corneometry Measurements During 12 Hours of Visit 2 | 0 hour, 2 hours, 4 hours, 6 hours, 8 hours and 12 hours (Visit 2)
  Six areas will be marked on the inner side of the participants' forearms, approximately 5 cm from the cubital region. These areas will be randomized, with 1 area for control (without product application) and the other 5 areas for product application, being each of them for 02 IPs (Facial Sunscreen A and Face Sunscreen B) and 3 benchmarks. The products will be applied topically only once in the marked areas. The 6 areas will be tested in triplicate at each experimental time (T0h, T2h, T4h, T6h, T8h and T12h) with the corneometer equipment.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielli Brianezi, Principal Investigator — Allergisa Pesquisa Dermato-Cosmética Ltda
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Consumer Inc. has an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu.
URL: http://yoda.yale.edu